CLINICAL TRIAL: NCT07036874
Title: Validation of Baveno VII Criteria and Spleen Stiffness Measurement on Outcome Prediction in Patients With Hepatocellular Carcinoma
Brief Title: Non-invasive Assessment for Outcome Prediction in Patients With Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jimmy Che-To Lai, Assistant Professor (Clinical), Chinese University of Hong Kong
Other Study IDs: 2024.249
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: HCC - Hepatocellular Carcinoma; Cirrhosis
Keywords: hepatocellular carcinoma; liver stiffness; spleen stiffness
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Store 10 mL of clotted blood and 10 mL of EDTA blood for future genetic and biochemical research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hepatocellular carcinoma: Adult patients with known chronic liver disease and hepatocellular carcinoma planning for curative-intent treatment
  Interventions: Diagnostic Test: transient elastography and oesophagogastroduodenoscopy

INTERVENTIONS:
Diagnostic Test: transient elastography and oesophagogastroduodenoscopy — Liver and spleen stiffness will be measured by transient elastography. Varices will be identified by oesophagogastroduodenoscopy.

SUMMARY:
This is a single-centre, prospective cohort study. Consecutive patients with compensated liver disease and hepatocellular carcinoma (HCC) for curative-intent treatment will be invited to this study. The study follow-up duration will be five years. The primary outcome is the composite of incident high-risk varices, hepatic decompensation and liver-related mortality. The participants will undergo transient elastography at baseline and then half-yearly post-HCC curative treatment; and oesophagogastroduodenoscopy (OGD) at baseline and then at year 1, 3 and 5 post-HCC curative treatment. Clinical assessments and laboratory tests will also be done at baseline and every 6 months until year 5 to identify any clinical events.

DETAILED DESCRIPTION:
1.1 Significance of chronic liver disease and hepatocellular carcinoma

Hepatocellular carcinoma (HCC) burdens the global healthcare system with a drastic increase in incidence by 70% from 1990 to approximately 747,000 cases and 480,000 deaths in 2019.

Despite implementation of screening ultrasound in at-risk populations and advances in the treatment of HCC in recent decades, HCC remains a lethal malignancy with a median survival of less than a year. Apart from the oncological factors, the underlying liver disease has an important impact on morbidity and mortality in patients with HCC as most HCC develop under the setting of chronic hepatic inflammation and fibrosis from patients with advanced chronic liver diseases of various aetiologies.

1.2 Non-invasive measurement of portal hypertension

In the Baveno VI consensus, the term "compensated advanced chronic liver disease" (cACLD) described spectrum of chronic liver diseases ranging from advanced liver fibrosis to compensated cirrhosis. Patients with cACLD are at risk of hepatic decompensation and development of HCC, especially for those with clinically significant portal hypertension (CSPH), which is conventionally measured invasively by hepatic venous pressure gradient (HVPG). The recently updated Baveno VII consensus implemented a non-invasive approach by incorporating liver stiffness measurement (LSM) by vibration-controlled transient elastography (VCTE) and platelet count in ruling in or out CSPH in patients with cACLD. In the Baveno VII consensus and as well incorporated into the latest practice guidance on portal hypertension, LSM ≤ 15kPa and platelet count ≥ 150 x 109/L rules out CSPH, whereas LSM > 25kPa, LSM 20-25kPa with platelet count <150 x 109/L or LSM 15-20kPa with platelet count <110 x 109/L rule in CSPH, prompting the presence of gastroesophageal varices. As well in Baveno VI consensus, LSM < 20 kPa with platelet count > 150 x 109/L also implies a minimal risk of high-risk varices and thus can have a screening oesophagogastroduodenoscopy (OGD) spared.

The development of spleen stiffness measurement (SSM) by VCTE also revolutionised the field by demonstrating its correlation with portal pressure and CSPH. Studies have shown that, by combining Baveno VII criteria with SSM, the accuracy in identifying CSPH (such as the presence of high-risk varices) was enhanced compared to adopting Baveno VII criteria alone.

1.3 Unmet need 1: Conflicting data on LSM/SSM in prediction of hepatic events in HCC patients

Use of LSM and SSM in prediction of HCC recurrence was reported in a few previous studies. The studies involved a one-stop LSM and/or SSM measurements with longitudinal follow-up on the recurrence rate of HCC. For instance, high baseline LSM was shown to be a poor prognostic factor in patients with HCC receiving radiofrequency ablation, and achieving low LSM reduced HCC recurrence. Another prospective study involving 175 patients with HCC suitable for resection showed that SSM was the only predictor for late HCC recurrence.

However, there are lack of data in the prediction of hepatic decompensation in patients with HCC. First, studies aiming to investigation on risk prediction of decompensation either excluded patients with HCC or regarded HCC as one of the study endpoints. Second, the present data available also showed conflicting results. For instance, two retrospective studies performed from our group suggested that Baveno VII criteria (i.e. LSM by VCTE and platelet count) could accurately identify high risk varices and hepatic events in both advanced HCC and that of different Barcelona Clinic Liver Cancer (BCLC) stages. On the contrary, another retrospective suggested that the use of both Baveno VI or VII criteria were inaccurate in predicting the presence of high-risk varices or CSPH measured by HVPG across different stages of HCC. Heterogeneity was present in the study subjects and data analysis among different studies, leading to divergent results. SSM as well was not included in these studies and that the effect of combined Baveno VII and SSM in prediction of decompensation in HCC patients is still uncertain.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Known chronic liver disease(s)
* HCC for curative-intent treatment (defined by HCC diagnosed with typical radiological features or histology, and planned for surgical resection or local ablative therapy as a curative-intent treatment)

Exclusion Criteria:

* Current or history of decompensated liver cirrhosis (i.e. Child's C cirrhosis, prior decompensating events such as ascites, variceal bleeding, hepatic encephalopathy and hepatorenal syndrome)

  o Child's B cirrhosis without decompensating events is not excluded
* Past history of HCC (ie. The current HCC is a recurrence of priorly treated HCC or a second de novo HCC after previous first HCC)
* Non-primary liver tumour (such as secondary liver tumour due to metastasis from another distant primary tumour)
* History of liver transplantation or plan for liver transplantation as the modality of curative-intent HCC treatment
* Asplenism or history of splenectomy
* Contraindication to OGD (eg. Intestinal perforation of obstruction)
* Serious medical illness with limited life expectancy of less than 6 months
* Pregnancy
* Unable to obtain or refusal of informed consent from patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients with hepatocellular carcinoma fulfilling the inclusion and exclusion criteria will be invited to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Composite of incident high-risk varices, hepatic decompensation and liver-related mortality | 5 years
  Composite of incident high-risk varices, hepatic decompensation and liver-related mortality

SECONDARY OUTCOMES:
Development of each hepatic decompensation event | 5 years
  Development of each hepatic decompensation event
Recurrence of hepatocellular carcinoma | 5 years
  Recurrence of hepatocellular carcinoma
Changes in Child-Pugh and Model for End-stage Liver Disease scores | 5 years
  The minimum and maximum Child-Pugh score are 5 and 15, respectively. The minimum and maximum Model for End-stage Liver Disease score are 6 and 40, respectively. A higher score denotes worse outcome in both score.
Change in liver and spleen stiffness measurements | 5 years
  Change in LSM and SSM

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy CT Lai, MB ChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after the first publication until 15 years after the end of the study
Access Criteria: By email communication

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT07036874/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT07036874/ICF_001.pdf